CLINICAL TRIAL: NCT03153462
Title: A Multicenter, Open-label, Expanded Access Study of Axicabtagene Ciloleucel for the Treatment of Subjects With Relapsed/Refractory Large B-cell Lymphoma.
Brief Title: Axicabtagene Ciloleucel Expanded Access Study
Acronym: ZUMA-9
Status: Approved for marketing | Type: Expanded Access
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Other Study IDs: KTE-C19-109; 2015-005007-86 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Relapsed/Refractory Diffuse Large B Cell Lymphoma; Relapsed/Refractory Primary Mediastinal B Cell Lymphoma; Relapsed/Refractory Transformed Follicular Lymphoma; Relapsed/Refractory High-Grade B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — axicabtagene ciloleucel

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — Axicabtagene Ciloleucel and A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by a single infusion of CAR transduced autologous T cells administered intravenously.
  Other Names: Yescarta®

SUMMARY:
A multicenter, open-label expanded access protocol for the treatment of subjects with relapsed/refractory large B-cell lymphoma.

Subjects who received an infusion of axicabtagene ciloleucel will complete the remainder of the 15 year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed large B-cell lymphoma, including the following types:

   1. DLBCL, not otherwise specified
   2. Primary mediastinal large B-cell lymphoma
   3. High-grade B-cell lymphoma
   4. DLBCL arising from follicular lymphoma (transformed follicular lymphoma, or TFL)
2. Relapsed or refractory disease, defined as one or more of the following:

   1. No response to first-line therapy (primary refractory disease); subjects who are intolerant to first-line therapy chemotherapy are excluded OR
   2. No response or relapse to second or greater lines of therapy OR
   3. Relapsed after ASCT
3. Subjects must have received adequate prior therapy including at a minimum:

   1. anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20 negative, and
   2. an anthracycline containing chemotherapy regimen;
4. No evidence, suspicion, and/or history of central nervous system (CNS) involvement of lymphoma
5. Age 18 or older
6. Eastern cooperative oncology group (ECOG) performance status of 0 or 1
7. Absolute neutrophil count ANC ≥1000/μL
8. Platelet count ≥75,000/μL
9. Absolute lymphocyte count ≥100/μL
10. Adequate renal, hepatic, pulmonary and cardiac function defined as:

    1. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min
    2. Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤2.5 upper limit of normal (ULN)
    3. Total bilirubin ≤1.5 mg/dL, except in subjects with Gilbert's syndrome.
    4. Cardiac ejection fraction ≥ 50% and no evidence of pericardial effusion within 180 days provide the subject did not receive an anthracycline based treatment or experience a cardiac event or change in performance status
    5. No clinically significant pleural effusion
    6. Baseline oxygen saturation >92% on room air
11. Cohort 2 inclusion criteria: Subjects whose commercial manufacture of axicabtagene ciloleucel did not meet commercial release specification(s)

Exclusion Criteria:

1. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years
2. History of allogeneic stem cell transplantation (SCT)
3. Prior CD19 targeted therapy
4. Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy
5. History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
6. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment and after consultation with the Kite Pharma Medical Monitor
7. History of human immunodeficiency virus (HIV) infection or acute or chronic active hepatitis B or hepatitis C infection. Subjects with a history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines
8. History or presence of primary CNS lymphoma and/or CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
9. Cohort 2 exclusion criteria: Any medical condition that, deemed by the investigator, may interfere with assessment of safety or efficacy of study treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (15):
- United States (15):
  - City of Hope, Duarte, California
  - Stanford Cancer Institute, Stanford, California
  - University of Miami Hospital and Clinics, Miami, Florida
  - H. Lee Moffitt Cancer and Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - The University of Kansas Hospital Investigational Drug Services, Westwood, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03153462